CLINICAL TRIAL: NCT05647694
Title: V-NAV: Advanced Indoor Navigation Aid for Individuals With Visual Impairments, End User Evaluation
Brief Title: V-NAV Usability Study: End Users Trying the Vortant Indoor Navigation Tool
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Usability issues were identified with the app. Some usability enhancements are being implemented prior to continuing with the study
Sponsor: Vortant Technologies, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NEI-VNAV-2C
Record Dates: First submitted 2022-11-29; First posted 2022-12-12 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Blindness and Low Vision
Keywords: blindness, indoor navigation
MeSH Terms: conditions — Blindness; Vision, Low

STUDY DESIGN:
Intervention Model Description: Participants will compare the value of the prototype app to their previous navigational experience without the app.
Masking Description: The use of the app will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-NAV users (Experimental): Users who try the V-NAV for navigation tasks.
  Interventions: Other: V-NAV indoor navigation prototype

INTERVENTIONS:
Other: V-NAV indoor navigation prototype — Users will use the V-NAV prototype as an augmentation to their indoor navigation activities.

SUMMARY:
The study will begin with an explanatory/training session where individuals with low vision will learn to use the V-NAV (Vortant NAVigation tool) indoor navigation app, and will have the opportunity to try it for a few representative tasks. The main activity includes a take-home trial, an extended unstructured period to emulate the post-purchase experience of users, during which participants will have the opportunity to use the V-NAV in their everyday lives. Data will be collected from the users to measure the relative advantage of V-NAV compared to the user's current indoor navigation method.

DETAILED DESCRIPTION:
The introductory session, emphasizing real-world experiences, will involve a brief training session followed by simulated navigation experiences in a convenient location to the users. Participants will use V-NAV to record approximately 8 locations, then will be given instructions to find these locations again. The V-NAV prototype's logging software will measure distance walked and task time. Participants will complete a study-specific tool covering the relevant attributes of the V-NAV prototype, as well as a standardized tool, the NASA TLX (Task Load Index).

Subsequently, participants will complete a take-home trial, during which they will be encouraged to use the V-NAV features regularly to support their everyday community navigation activities. Participants will be contacted approximately weekly with a "check-in" to answer questions and resolve any emergent technical problems. At the conclusion of the trial, a product-specific tool and an appropriate standardized tool, the PIADS (Psychosocial Impact of Assistive Devices Scale) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* AFB "visually impaired" definition, acuity 20/70 or worse or field loss of 140 degrees

Exclusion Criteria:

* Any health condition that may affect safety of individual to participate
* Any physical, mental, or behavioral impairment that would provide more than minimal risk or hindering ability to comprehend the purpose of the device or otherwise to be a potential user of the V-NAV hardware or app.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
V-NAV effectiveness | 4 weeks
  A measurement of user impressions as to the value of the V-NAV navigation aid. Use of e.g., PIADS survey.

SECONDARY OUTCOMES:
V-NAV usability | 1 day
  A measurement of how usable the V-NAV is. Use of e.g., NASA TLX survey.

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Schaefer, M.S.E, Principal Investigator — Vortant Technologies, LLC
Locations (1):
- Vortant Technologies, Weaverville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No